CLINICAL TRIAL: NCT00885950
Title: Prevention of the Hepatic Sinusoidal Obstruction Syndrome Secondary to Oxaliplatin-based Neoadjuvant Chemotherapy for Colorectal Liver Metastases by Means of Anticoagulants
Brief Title: Prevention of the Hepatic Sinusoidal Obstruction Syndrome by Means of Anticoagulants
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-4-076
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Sinusoidal Obstruction Syndrome; Colorectal Liver Metastases
Keywords: colorectal liver metastases; neoadjuvant chemotherapy; oxaliplatin; sinusoidal obstruction syndrome; anticoagulants
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin embedded liver tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colorectal liver metastases: Patients with colorectal liver metastases undergoing partial hepatic resection who were preoperatively treated with either neoadjuvant chemotherapy or not and/or anticoagulants or not

SUMMARY:
The purpose of the study is to determine whether anticoagulant use (i.e. salicylates, clopidogrel, low-molecular weight heparin, or coumarin derivates) is able to prevent the development of the sinusoidal obstruction syndrome secondary to oxaliplatin-based neoadjuvant chemotherapy in patients suffering from colorectal liver metastases.

DETAILED DESCRIPTION:
Surgical resection remains the only curative treatment for patients suffering from colorectal liver metastases, but only 15-25% of patients are initially eligible for resection. The majority of patients suffering from colorectal liver metastases receives chemotherapy prior to liver surgery in order to downsize the colorectal liver metastases. Preoperative treatment with oxaliplatin-based chemotherapy is related to sinusoidal injury, the so-called sinusoidal obstruction syndrome. Patients with histologically proven sinusoidal injury undergoing liver surgery have a higher risk of post-resectional morbidity. Damage to the hepatic sinusoids is a key factor for the development of the sinusoidal obstruction syndrome. Anticoagulants (i.e. salicylates, clopidogrel, low-molecular weight heparin, or coumarin derivates) might be able to prevent this damage and, consequently, the development of the sinusoidal obstruction syndrome in patients suffering from colorectal liver metastases treated with neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* colorectal liver metastases that are eligible for resection
* operated from January 2008 up until December 2009 at Maastricht University Medical Centre

Exclusion Criteria:

* irresectable colorectal liver metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from colorectal liver metastases who have undergone a partial hepatic resection
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Histologically proven hepatic sinusoidal injury | during liver surgery

SECONDARY OUTCOMES:
90-day morbidity and mortality | up until 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven WM Olde Damink, MD, PhD, MSc, Principal Investigator — Maastricht University Medical Centre; Rob Jansen, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Department of Surgery; Maastricht University Medical Centre, Maastricht, Netherlands